CLINICAL TRIAL: NCT03825120
Title: The Longitudinal Evaluation of Ovarian Aging and Cardiovascular Risk
Acronym: OVACV
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AG053332 (NIH); 1R01AG053332-01A1 (NIH)
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infertility; Cardiovascular Risk Factor
Keywords: reproductive health; fertility; infertility; aging; health; cardiovascular disease; cardiovascular disease risk
MeSH Terms: conditions — Infertility; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women from original OVA cohort

SUMMARY:
Despite significant improvements in prevention and treatment of cardiovascular disease (CVD), the growing aging population suggests CVD will continue to pose a significant public health burden. Women are a special group where microvascular disease is more common and traditional risk factors may not fully identify risk. Women's reproductive history (e.g. menarcheal age, menstrual cycles, infertility, pregnancy, menopause) may pose unique risk and suggests an opportunity for new approaches. The investigators propose a women-centered approach for early identification of women at risk that investigates the unique loss of reproductive function at an age long before other vital systems fail. Despite its importance, little is known about the determinants or correlates of ovarian aging, or the health implications, especially in diverse communities. Only recently have reliable biomarkers of the remaining oocyte pool been available for use in normally cycling women. This availability gives us a unique opportunity to characterize the association between "ovarian age" (cross-sectional) and the rate of "ovarian aging" or oocyte decline over time (longitudinal) and the health implications of accelerated oocyte loss. The investigators hypothesize ovarian age/aging provides a window onto the general health of women. The investigators suggest it is not the progressive deficiency of estrogen with menopause that increases risk, but common underlying cellular aging mechanisms first evident in young populations as lower ovarian reserve (follicle number) due to the unique sensitivity of the ovary.

Studies of cellular aging focused on mitochondrial dysfunction, oxidative stress, inflammation, and telomere length have identified correlations with CVD risk. Improved understanding of the mechanisms of cellular aging suggests telomere shortening and dysfunction may drive mitochondrial dysfunction and potentially the parallel between cellular aging and CVD. The oocyte is particularly sensitive to mitochondrial dysfunction, having 10 times the number of mitochondria as any somatic cell. Additionally, mitochondrial dysfunction and telomere shortening have been associated with ovarian aging. This begs the question of whether, given the susceptibility of the ovary to mitochondrial dysfunction, accelerated ovarian aging may be a harbinger of subsequent CVD risk. To address this critical question, the investigators propose to leverage the largest and most ethnically diverse population of normal reproductive-aged women, with detailed measures of ovarian age, and to deploy peripheral endothelial function testing, a non-invasive sensitive marker of early CVD risk. Ovarian aging is thought to be largely genetically determined, but the impact of race/ethnicity has not been fully explored. Evaluating the impact of ethnicity on ovarian aging, and combining this information with the impact of modifiable behavioral risk factors, may help clarify CVD risk in young, ethnically-diverse, reproductive-age women. The investigators believe improving our understanding of factors that affect the rate of oocyte/follicle loss and the relationship with CVD risk factors will promote a novel method to identify women at earlier and/or increased cardiac risk.

DETAILED DESCRIPTION:
The investigators propose to carry out three Specific Aims:

1. Determine whether markers of ovarian age/aging are associated with increased CVD risk.

   Specifically, the investigators propose to assess whether:
   1. Ovarian age predicts CVD risk (measured by peripheral endothelial function testing) independent of chronological age.
   2. The rate of ovarian aging is independently associated with increased CVD risk after adjustment for ovarian and chronological age.
2. Determine whether ovarian aging may moderate or mediate established associations between race/ethnicity and CVD risk and socio/emotional health and CVD risk. Specifically, the investigators propose to:

   1. Examine whether observed race/ethnic disparities in CVD risk (measured by peripheral endothelial function testing) may vary by (moderation model) or be partially attributable to (mediation model) ovarian aging.
   2. Examine whether effects of socio/emotional health (as indexed by separate composites of psychosocial functioning and socioeconomic status) on CVD risk may vary by (moderation model) or be partially attributable to (mediation model) ovarian aging.
3. Determine if similar mechanisms of cellular aging underlie both ovarian aging and CVD risk. Temporal appearance of indices of cellular aging, ovarian aging and CVD risk would support our primary hypothesis. Specifically, we propose to determine whether telomere and mtDNA in peripheral leukocytes, oxidative stress (plasma F2-isoprostanes), and indices of inflammation (C-reactive protein, interleukin-6, and soluble intercellular adhesion molecule-1) correlate with both ovarian aging and CVD risk, and the temporal pattern of appearance.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment into the original OVA cohort (NCT00501800)

Exclusion Criteria:

* Not a member of the original OVA cohort

Ages: 35 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: * member of Northern California Kaiser Permanente Health Plan at time of enrollment into original OVA cohort
  * self-identifying as Caucasian, Chinese, Filipino, African-American, or Hispanice (Mexican or Central American)
Sampling Method: Non-Probability Sample
Enrollment: 865 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Change in the EndoScore or reactive hyperemia ratio, an index of peripheral endothelial function, as assessed by the FDA-approved EndoPAT 2000 | 2 times, once at each of 2 study visits ~1 year apart
  Endothelium-mediated changes in vascular tone will be represented by the EndoScore or ratio of Reactive Hyperemia pre-occlusion to post-occlusion of the brachial artery (via blood pressure cuff). A score > 1.67 is considered "normal" and a score <= 1.67 is "abnormal". The EndoPAT 2000 machine will be used for this measure, which is the only non-invasive method of measuring endothelial function or the state of arterial health. Well-functioning arteries protect blood vessels from hardening (or atherosclerosis) and plaque build up. The EndoScore score will be the primary measure for cardiovascular (CV) disease risk, as actual CV event rates will be too low for many years

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle I Cedars, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No